CLINICAL TRIAL: NCT05756582
Title: Cross-sectional Study on Prevalence of Latent Tuberculosis Infection in Health-care Workers and Students. A GENERATOR Infrastructure.
Brief Title: Prevalence of Latent Tuberculosis Infection in Health-care Workers and Students
Acronym: CROSSWORD
Status: Recruiting | Type: Observational
Sponsor: Eleonora Nucera (Other)
Responsible Party: Sponsor-Investigator, Eleonora Nucera, Head of Allergy Unit, Catholic University of the Sacred Heart
Organization: Catholic University of the Sacred Heart (Other)
Other Study IDs: ID3528
Record Dates: First submitted 2023-02-19; First posted 2023-03-06 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Tuberculosis; Tuberculosis, Pulmonary; Tuberculosis Infection; Latent Tuberculosis; Health Care Associated Infection
Keywords: latent tuberculosis infection; health-care workers; students; survey
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary; Latent Tuberculosis; Cross Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health-care workers and students: The study will involve all health-care workers of Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome - a tertiary reference hospital with over 1,500 beds - and all students of all three-year and single-cycle degree courses, master's degree courses, graduate schools of the faculty of Medicine and Surgery of the Catholic University of Sacred Heart in Rome, trained at the Fondazione Policlinico Universitario A. Gemelli IRCCS.
  Interventions: Diagnostic Test: Prevalence of Latent Tuberculosis Infection

INTERVENTIONS:
Diagnostic Test: Prevalence of Latent Tuberculosis Infection — The prevalence of Latent Tuberculosis Infection [LTBI] is defined as 1) tuberculin conversion after a documented negative-baseline tuberculin skin test (TST), 2) positive result of the QuantiFERON-TB Gold (QFT) test performed [higher response than the cut-off value of 0.35 IU / ml of INF-γ was detected in at least one test tube (TB1 or TB2)], 3) chest imaging excluding pleural and/or pulmonary lesions suggestive of active tuberculosis and 4) final medical evaluation done by a Specialist in Infectious Diseases which excluded active disease. All four criteria must be met.

SUMMARY:
This study is a cross-sectional study that examines the prevalence of Latent Tuberculosis Infection [LTBI], defined as individuals infected with Mycobacterium tuberculosis with no clinical evidence of disease, and the possible risk factors of LTBI in a large cohort of health care workers (HCWs) and students.

DETAILED DESCRIPTION:
Mycobacterium tuberculosis may develop symptoms and signs of disease or may have no clinical evidence of disease (latent tuberculosis infection [LTBI]). TB disease remains one of the major causes of morbidity and mortality in the world.

A survey to assess the prevalence of the individuals with a LTBI and evaluate the potential main risk-factors will be performed on both HCWs and students attending the hospital wards, trained at Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome.

This study is a cross-sectional study that examines the prevalence of Latent Tuberculosis Infection [LTBI], defined as individuals infected with Mycobacterium tuberculosis (MT) with no clinical evidence of disease, and the possible risk factors of LTBI in a large cohort of health care workers (HCWs) and students.

The study will involve all HCWs of Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome - a tertiary reference hospital with over 1,500 beds - and all students of all three-year and single-cycle degree courses, master's degree courses, graduate schools of the faculty of Medicine and Surgery of the Catholic University of Sacred Heart in Rome, trained at the Fondazione Policlinico Universitario A. Gemelli IRCCS.

All enrolled participants, who will agree to participate to the study and answer the questionnaire, will respond a cross-sectional questionnaire survey through dedicated tablet. The survey will contain a brief explanation of the study aims and an invitation to respond to a 9 items multiple choice questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* all health-care workers of Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome,
* all students of all three-year and single-cycle degree courses, master's degree courses, graduate schools of the faculty of Medicine and Surgery of the Catholic University of Sacred Heart in Rome, trained at the Fondazione Policlinico Universitario A. Gemelli IRCCS,
* written informed consent.

Exclusion Criteria:

* denied informed consent.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will involve all HCWs of Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome - a tertiary reference hospital with over 1,500 beds - and all students of all three-year and single-cycle degree courses, master's degree courses, graduate schools of the faculty of Medicine and Surgery of the Catholic University of Sacred Heart in Rome, trained at the Fondazione Policlinico Universitario A. Gemelli IRCCS.
Sampling Method: Probability Sample
Enrollment: 2040 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
The prevalence of Latent Tuberculosis Infection | At enrollment.
  The prevalence of Latent Tuberculosis Infection [LTBI] defined as 1) tuberculin conversion after a documented negative-baseline tuberculin skin test (TST), 2) positive result of the QuantiFERON-TB Gold (QFT) test performed [higher response than the cut-off value of 0.35 IU / ml of INF-γ was detected in at least one test tube (TB1 or TB2)], 3) chest imaging excluding pleural and/or pulmonary lesions suggestive of active tuberculosis and 4) final medical evaluation done by a Specialist in Infectious Diseases which excluded active disease. All four criteria must be met.

SECONDARY OUTCOMES:
Age | At enrollment.
  Age as possible risk factor of Latent Tuberculosis Infection.
Sex | At enrollment.
  Sex as possible risk factor of Latent Tuberculosis Infection.
Vaccination history | At enrollment.
  Bacillus Calmette-Guérin (BCG) vaccination history as possible risk factor of Latent Tuberculosis Infection.
Previous work or stay in other at risk countries | At enrollment.
  Previous work or stay in other countries with high TB rates including Armenia, Azerbaijan, Belarus, Bulgaria, Estonia, Georgia, Kazakhstan, Kyrgyzstan, Latvia, Lithuania, Moldova, Romania, Russia, Tajikistan, Turkey, Turkmenistan, Ukraine and Uzbekistan; as possible risk factor of Latent Tuberculosis Infection.
Recent exposure | At enrollment.
  Known recent (within 6 months) exposure to TB-infected patient; as possible risk factor of Latent Tuberculosis Infection.
Smoking | At enrollment.
  Current smoking as possible risk factor of Latent Tuberculosis Infection.
Co-morbidities / medical history | At enrollment.
  Co-morbidities / medical history [HIV, diabetes, silicosis, chronic kidney disease, solid organ transplant, malignant hematologic malignancies or undergoing chemotherapy, gastrectomy or fasting bypass, biological drugs]; as possible risk factor of Latent Tuberculosis Infection.
QuantiFERON-TB | At enrollment.
  Median QuantiFERON-TB Gold In-Tube level (TB Ag-Nil) as possible risk factor of Latent Tuberculosis Infection.
Occupation | At enrollment.
  Occupation [doctor, nurse, laboratory technicians, paramedical personnel, "preclinical" students with no contact with patients inside the hospital, and "clinical" students attending various medical, laboratory, and surgical departments of the hospital, including the infectious disease wards] as possible risk factor of Latent Tuberculosis Infection.
Working / training Unit | At enrollment.
  Working / training Unit as possible risk factor of Latent Tuberculosis Infection.
Years working as HCW | At enrollment.
  Years working as HCW as possible risk factor of Latent Tuberculosis Infection.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Rizzi, MD, PhD, Principal Investigator — Catholic University of Sacred Heart; Eleonora G Nucera, Prof., MD, Principal Investigator — Catholic University of Sacred Heart; Domenico Staiti, Prof., MD, Principal Investigator — Catholic University of Sacred Heart; Antonio Gasbarrini, Prof., MD, Study Director — Catholic University of Sacred Heart; Vincenzo Valentini, Prof., MD, Study Director — Catholic University of Sacred Heart
Locations (1):
- UOSD Allergologia e Immunologia Clinica, Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

REFERENCES:
- [Derived] Rizzi A, Nucera E, Mazzucco W, Palumbo P, Staiti D, Moscato U, De Simone FM, Sali M, Boldrini L, Capocchiano ND, Patarnello S, Rumi G, Chini R, Carusi V, Centrone M, Di Rienzo A, Longhino D, Laface C, Mellone S, Maida CM, Cannizzaro E, Cirrincione L, Verso MG, Saracino A, Di Gennaro F, Vimercati L, De Maria L, Sponselli S, Scoppettuolo G, Pastorino R, Gasbarrini A, Inchingolo R. An interoperable web-based platform to support health surveillance against latent tuberculosis infection in health care workers and students: The evolution of CROSSWORD study protocol. PLoS One. 2025 Mar 25;20(3):e0319568. doi: 10.1371/journal.pone.0319568. eCollection 2025. PMID 40132007